CLINICAL TRIAL: NCT03482206
Title: Automated Extracranial Internal Carotid Artery Ultrasound Sensor for Traumatic Brain Injury
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Need more time to optimize the sensor
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Cindy Hsu, Assistant Professor, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HUM00137659
Record Dates: First submitted 2018-03-20; First posted 2018-03-29 (Actual); Last update posted 2019-08-19 (Actual); Status verified 2019-08

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy subjects (Experimental): Healthy adult volunteers (age 18 or greater) that are not claustrophobic, do not have hyperventilation or panic disorders, not pregnant, have no metal implants and can pass the MRI screening questions.
  Interventions: Device: Automated extracranial internal carotid artery ultrasound sensor

INTERVENTIONS:
Device: Automated extracranial internal carotid artery ultrasound sensor — The investigators' goal is to develop a wearable noninvasive, continuous, automated ultrasound sensor to accurately measure arterial blood flow volume outside of the head. Ultrasound uses sound waves to create a picture. In doing so, the investigators hope to detect CBF compromise early, preventing secondary injuries in TBI patients.

SUMMARY:
Traumatic brain injury (TBI) affects 1.7 million people in the United States each year, resulting in 2.5 million emergency department visits, 280,000 hospitalizations, >50,000 deaths, and more than $60 billion in economic cost. TBI also affects >30,000 military personnel annually and almost 8% of veterans who received care between 2001 and 2011. Post-traumatic neurologic outcome depends on the severity of initial injuries and the extent of secondary cerebral damage. Ischemia is the most common and devastating secondary insult. Ischemic brain damage has been identified histologically in ~90% of patients who died following closed head injury, and several studies have associated low cerebral blood flow (CBF) with poor outcome. Specifically, CBF of less than 200 ml/min has been shown to be the critical lower threshold for survival in neurointensive care patients. In addition to intracranial hypertension and cerebral edema, systemic hypotension and reduced cardiac output contribute substantially to posttraumatic cerebral ischemia. Additionally, the carotid artery is the most common site of blunt cerebral vascular injury (BCVI), which may further compromise CBF and cause subsequent death or debilitating stroke. Specifically, high grade internal carotid arterial (ICA) injuries are associated with the highest mortality and stroke rate.

The investigators' goal is to develop of a wearable noninvasive, continuous, automated ultrasound sensor to accurately measure extracranial ICA flow volume. In doing so, the investigators aim to enable early detection of CBF compromise, thereby preventing secondary ischemic injuries in TBI patients. To achieve this goal, the investigators plan to first build a prototype wearable ICA ultrasound senor with integrated signal processing platform, then test its accuracy in an in vitro system and healthy human subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Age 18 or older

Exclusion Criteria:

* Claustrophobic
* Hyperventilation or panic disorders
* Pregnant
* Have metal implants or cannot pass the MRI screening questions

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Internal carotid artery blood flow | 5 minutes before ultrasound or MRI measurement until 15 minutes after the measurement
  The investigators will measure volume of blood flow through the extracranial internal carotid artery using the ultrasound sensor and MRI

SECONDARY OUTCOMES:
End tidal CO2 level | 5 minutes before ultrasound or MRI measurement until 15 minutes after the measurement
  End tidal carbon dioxide level during normal, hypoventilation, and hyperventilation

IPD SHARING:
Plan to Share IPD: No